CLINICAL TRIAL: NCT06315829
Title: A Machine Learning Approach to Infantile Spasms Recognition in Video Recordings
Brief Title: Artificial Intelligence-based Video Analysis to Detect Infantile Spasms
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00429753
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Infantile Spasms
Keywords: Seizure; Epilepsy; Infantile Spasm; Epileptic Spasm; West Syndrome; Hypsarrhythmia; Artificial Intelligence; Video Analysis; Computer Vision; Machine Learning
MeSH Terms: conditions — Spasms, Infantile; Seizures; Epilepsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Confirmed Epileptic Spasms (Positive Class): Participants diagnosed with infantile spasms based upon historical data and supportive electroencephalography data (i.e. hypsarrhythmia or modified hypsarrhythmia background).
  Interventions: Device: Spasm Vision
- Epileptic Spasm Mimics (Negative Class): Participants diagnosed with non-epileptic movements (e.g. Sandifer syndrome, shuddering attacks, stretching, stereotypy, startle reflex, writhing movements, jitteriness, sleep myoclonus) based upon historical data and supportive electroencephalography data (when available).
  Interventions: Device: Spasm Vision
- Awake and Alert (Negative Class): Participants exhibiting spontaneous, subtle movements in the awake and alert state.
  Interventions: Device: Spasm Vision

INTERVENTIONS:
Device: Spasm Vision — Machine learning software developed to analyze videos and accurately distinguish infantile spasms from visually similar movements.

SUMMARY:
Infantile spasms are a type of seizure linked to developmental issues. Unfortunately, they are often misdiagnosed, causing delays in treatment. The purpose of this study is to develop a computer program that can reliably differentiate infantile spasms from similar, yet benign movements in videos. This computer program will learn from videos taken by parents of study participants. Quickly recognizing and treating infantile spasms is crucial for ensuring the best developmental outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participant age less than 24 months
* Participant evaluated in the Johns Hopkins Outpatient Center, Johns Hopkins Pediatric Emergency Department or Johns Hopkins Inpatient Units due to spells of abnormal movement or seizure
* Participant evaluated by a pediatric neurologist during the outpatient or inpatient visit at Johns Hopkins Hospital
* At least one video recording of the spell of abnormal movement produced by the parent/guardian available for provider review

Exclusion Criteria:

* Poor video recording quality
* Entire patient is not in frame

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants will be recruited from the outpatient and inpatient settings of Johns Hopkins Hospital, an academic medical center located in Baltimore, Maryland offering tertiary and quaternary care.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Model Sensitivity (Recall) | 2 years
  Proportion of true positives which the model classified correctly in the test dataset.
Model Specificity | 2 years
  Proportion of true negatives which the model classified correctly in the test dataset.
Model Positive Predictive Value (Precision) | 2 years
  Proportion of positive classifications which were correct in the test dataset.
Model Negative Predictive Value | 2 years
  Proportion of negative classifications which were correct in the test dataset.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Kossoff, MD, Principal Investigator — Johns Hopkins Neurology; Rama Chellappa, PhD, Principal Investigator — Johns Hopkins Biomedical Engineering
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No